CLINICAL TRIAL: NCT01448343
Title: Effect of Rapid Transfusion With FMS(Fluid Management System 2000®) on the Plasma Potassium Concentration in Adult Liver Transplantation Recipients)
Brief Title: Effect of Rapid Transfusion With Fluid Management System 2000® (FMS)
Acronym: FMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CWJung_FMS
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Liver Transplantation
Keywords: transfusion; potassium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FMS (Experimental): Patients who received blood transfusion using FMS
  Interventions: Device: Fluid management system 2000 (FMS)

INTERVENTIONS:
Device: Fluid management system 2000 (FMS) — The FMS has an integrated large volume (about 3000 ml) reservoir and delivers a blood mixture (4 unit RBC, 4 unit FFP and 800 ml normal saline) put in the reservoir at a maximum rate of 750 ml/min.

SUMMARY:
Rapid infusion of red blood cells is known to result in the increase of plasma potassium. The researchers are trying to investigate the change in plasma potassium during rapid infusion of mixed blood components in the reservoir of the fluid management system (FMS) in liver transplant recipients.

DETAILED DESCRIPTION:
FMS is a standard equipment to prepare for the massive bleeding during the liver transplant surgery. This device usually delivers a mixture of red blood cell (RBC), fresh frozen plasma and normal saline. Rapid infusion of RBC is known to result in the increase of potassium and the decrease of calcium in the plasma of the patient. However there is no report about the consequence of rapid transfusion of the blood mixture in the reservoir of the FMS, especially in the liver transplantation recipients. The primary end point of this study is to investigate the change in the plasma potassium and to assess the possibility of hyperkalemia and related morbidity. Changes of blood pH and plasma calcium will also be sought.

ELIGIBILITY:
Inclusion Criteria:

* liver transplantation recipients

Exclusion Criteria:

* hemoglobin > 10 g/dL before surgery
* renal failure
* hyperkalemia
* chronic hyponatremia
* cardiac dysfunction

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Plasma potassium | Transfusion and sampling of blood are made intraoperatively, mainly during the period of hepatectomy. Overall time of data collection is usually within 4 hrs.
  Four units of RBC, four units of FFP and 800 ml of normal saline are put into the FMS reservoir. Samplings of blood are made before, during and after the transfusion of 300 ml of blood mixture. Sites of blood samplings are the infusion line of the FMS and the arterial and central venous lines of the patient. This process is repeated 4 times in a patient. Acquired blood samples are immediately analyzed with a point of care test device (GEM Premier 3000). The result will be analyzed with appropriate statistics such as RMANOVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea